CLINICAL TRIAL: NCT04196907
Title: Noninvasive Hemoglobin Spot Check Repeatability and Reproducibility in a Blood Donation Setting
Brief Title: Rad-67 Repeatability and Reproducibility
Status: Completed | Type: Interventional
Sponsor: Masimo Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SDBB0002
Record Dates: First submitted 2019-12-03; First posted 2019-12-12 (Actual); Results first posted 2021-09-29 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Unapproved Device: Yes

ARMS (1):
- Test subjects (Experimental): All subjects are enrolled and receive Rad-67 Pulse Oximeter and DCI Mini sensor for measurement of hemoglobin.
  Interventions: Device: Rad-67 Pulse CO-Oximeter and DCI Mini sensor

INTERVENTIONS:
Device: Rad-67 Pulse CO-Oximeter and DCI Mini sensor — Noninvasive Pulse CO-Oximeter device and sensor are used to measure hemoglobin.

SUMMARY:
The primary objective of this clinical investigation is to evaluate the repeatability and reproducibility of using Rad-67 Pulse CO-Oximeter

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Weight at least 110 pounds
* Subjects with the intention of being screened for eligibility to donate blood
* The subject has given written informed consent to participate in the study

Exclusion Criteria:

* Subjects with skin abnormalities at the planned application sites that may interfere with sensor application, per directions-for-use (DFU) or trans-illumination of the site, such as burns, scar tissue, infections, abnormalities, etc.
* Subjects unwilling to remove nail polish or acrylic nails
* Subjects with blood cancers such as leukemia
* Subjects with hemoglobin disorders such as sickle-cell anemia and thalassemia or with known history of infectious diseases such as HIV/AIDS, syphilis, hepatitis, etc.
* Subjects with self-disclosed/known pregnancy at the time of enrollment
* Subjects deemed not suitable for the study at the discretion of the investigator
* Subjects unlikely to be able to refrain from excessive motion during data collection. Excessive motion includes postural changes, making hand gestures, involuntary muscular movements, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-11-19 (Actual); Primary Completion 2019-11-20 (Actual); Study Completion 2019-11-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- San Diego Blood Bank, San Diego, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Test Subjects
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Test Subjects
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 19
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 11
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 0
  White | 8
  More Than One Race | 0
  Unknown or Not Reported | 0
  Hispanic | 9
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Variation Ratio of Total Repeatability and Reproducibility Hemoglobin Measurements Using Rad-67.
Description: Quality of hemoglobin measurements is defined as a variance ratio of total Gage repeatability and reproducibility variance to total variance. Subject, operator and device were considered as components to calculate this ratio.
Time Frame: 1 hour
Measure: Number; unit: ratio of variance
Arm/Group | Test Subjects
Number analyzed (Participants) | 20
ratio of variance | 10

ADVERSE EVENTS:
Time Frame: 1 hour
Arm/Group | Test Subjects
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-14): https://cdn.clinicaltrials.gov/large-docs/07/NCT04196907/Prot_SAP_000.pdf